CLINICAL TRIAL: NCT02342431
Title: Comparison of a Patient Warming System Using a Forced-air, Non-compressible Under-body Mattress Versus a Regular Forced-air Underbody Mattress System During Pediatric Cardiac Catheterization
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Cardiac Catheterization no longer part of the anesthesia department A (no belonging to cardiac anesthesia, which is a different department)
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Oliver Kimberger, Assoc.Prof PD Dr. MSc, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: momo_bh_1
Record Dates: First submitted 2012-11-13; First posted 2015-01-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Hypothermia
Keywords: Thermoregulation; Pediatric Anesthesia; Cardiac Catheterization
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Forced air compressible warming (Active Comparator): Warming with a compressible forced air mattress
  Interventions: Device: Forced air warming compressible
- Forced air non-compressible (Experimental): Warming with a non-compressible forced air mattress
  Interventions: Device: Forced air non-compressible

INTERVENTIONS:
Device: Forced air warming compressible — Warming with a compressible forced air mattress
  Arms: Forced air compressible warming
Device: Forced air non-compressible — Warming with a non-compressible forced air mattress
  Arms: Forced air non-compressible

SUMMARY:
The study is a comparison of a patient warming system using a forced-air, non-compressible under-body mattress (Möck & Möck, Hamburg, Germany) versus a regular forced-air underbody mattress system during pediatric cardiac catheterization in 40 patients.

The hypothesis is, that the non-compressible mattress provides better warming with less incidence of perioperative hypothermia (Core temperature < 36 °C) and faster warming slope (°C / time). The study is prospective, randomized, controlled and single-blinded.

Inclusion criteria will be pediatric patients < 1 year of age without fever or a treatment of therapeutic hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient scheduled for cardiac catheterization (diagnostic and/or interventional)< 1 year old

Exclusion Criteria:

* fever or therapeutic hypothermia

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypothermia | during surgery (1 - 6 hours)

SECONDARY OUTCOMES:
Core Temperature Slope | during surgery (1 - 6 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Kimberger, PD, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria